CLINICAL TRIAL: NCT05181683
Title: A Phase 1, Randomized, Open-Label Study Assessing the Safety and Tolerability of Co-Formulated Anti-Spike (S) SARS-CoV-2 Monoclonal Antibodies (Casirivimab+Imdevimab) in Adult Volunteers
Brief Title: COVID-19 Study Assessing the Safety and Tolerability of Co-Formulated Anti-Spike (S) SARS-CoV-2 Monoclonal Antibodies (Casirivimab+Imdevimab) in Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R10933-10987-COV-2179
Record Dates: First submitted 2022-01-04; First posted 2022-01-06 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Healthy; Chronic Stable Illness
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-COV-2)
MeSH Terms: conditions — COVID-19 | interventions — casirivimab and imdevimab drug combination; casirivimab; imdevimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Co-formulated casirivimab+imdevimab SC (Experimental): Randomized 1:1
  Interventions: Drug: Casirivimab+Imdevimab
- Co-formulated casirivimab+imdevimab IV (Experimental): Randomized 1:1
  Interventions: Drug: Casirivimab+Imdevimab

INTERVENTIONS:
Drug: Casirivimab+Imdevimab — Randomized 1:1 for intravenous (IV) or subcutaneous (SC) administration
  Other Names: REGN-COV2; Casirivimab; Imdevimab; REGEN-COV™; Ronapreve™

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of co-formulated subcutaneous (SC) and intravenous (IV) casirivimab+imdevimab

The secondary objectives of the study are to:

* Explore variability in the drug concentration profiles of casirivimab and imdevimab after co-formulated subcutaneous (SC) or intravenous (IV) administration
* Characterize the immunogenicity of casirivimab and imdevimab in serum over time

ELIGIBILITY:
Key Inclusion Criteria:

1. Is healthy, or has chronic medical condition(s) that per the opinion of the investigator is (are) stable, well-controlled, and not likely to require medical intervention through the end of study
2. Does not require medication(s) for co-morbid condition, or has received stable medication(s) for co-morbid condition(s) for at least 6 months prior to screening
3. Weighs between ≥60 kg and ≤100 kg at the time of screening
4. Has SARS-CoV-2-negative reverse-transcriptase polymerase chain reaction (RT-PCR) from a sample collected ≤72 hours prior to randomization, using local assay and sample collection and assay standards
5. Has completed a full course of COVID-19 vaccination more than 6 weeks prior to randomization

Key Exclusion Criteria:

1. Has active respiratory or non-respiratory symptoms consistent with COVID-19 in the opinion of the Investigator
2. Has recent SARS-CoV-2 infection that resolved within 6 weeks prior to randomization
3. Prior use of casirivimab+imdevimab at any time prior to randomization
4. Prior, current, or planned use during the study of any of the following treatments: COVID-19 convalescent plasma, other monoclonal antibodies against SARS-CoV-2 (eg, bamlanivimab and etesevimab, sotrovimab), intravenous immunoglobulin (any indication), or any other investigational, authorized, or approved agent intended for COVID-19 treatment or prevention (with the exception of COVID-19 vaccines)
5. Treatment with another investigational drug in the last 30 days or within 5 half-lives of the investigational drug, whichever is longer, prior to screening
6. Body mass index (BMI) ≥28 kg/m2
7. Medically-attended acute illness, systemic antibiotics use, or hospitalization for any reason within 30 days prior to screening
8. Acute exacerbation of a chronic pulmonary condition (eg, chronic obstructive pulmonary disease [COPD], asthma exacerbations) in the past 6 months prior to screening
9. Uncontrolled hypertension, in the opinion of the investigator
10. History of heart failure hospitalization, diagnosis of a myocardial infarction, stroke, transient ischemic attack, unstable angina, percutaneous or surgical revascularization procedure (coronary, carotid, or peripheral vascular), or intracardiac device placement (eg, pacemaker) within 12 months prior to screening
11. Cancer requiring treatment currently or in the past 5 years, except for non-melanoma skin cancer or cervical/anus in-situ
12. Is pregnant at screening

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Targeted grade ≥3 treatment-emergent adverse events (TEAEs) | Through end of study, approximately 16 weeks
Grade ≥3 injection-site reactions (ISRs) | Through end of study, approximately 16 weeks
Grade ≥2 infusion-related reactions (IRRs) | Through end of study, approximately 16 weeks
Grade ≥2 hypersensitivity reactions | Through end of study, approximately 16 weeks
Serious adverse events (SAEs) | Through end of study, approximately 16 weeks

SECONDARY OUTCOMES:
Concentrations of casirivimab and imdevimab in serum over time | Up to 16 weeks
Incidence and titer of anti-drug antibodies (ADA) to casirivimab and imdevimab | Up to 16 weeks
Incidence of neutralizing antibodies (NAb) to casirivimab and imdevimab | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Regeneron Study Site, Miami, Florida
  - Regeneron StudySite, Winter Park, Florida

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/